CLINICAL TRIAL: NCT06242340
Title: The Effect of Newborn's First Bath Time on Physiological Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, İlknur KAHRİMAN, Associate Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KARADENIZTEKNIK
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Baths
Keywords: infant, intensive care unit, baths, touch

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Preterm (between 32 0/7 and 36 6/7 weeks)
  Interventions: Other: Preterm group bathing 24 hours after birth.
- Group 2 (Experimental): Preterm (between 32 0/7 and 36 6/7 weeks)
  Interventions: Other: Preterm group bathing 48 hours after birth.
- Group 3 (Experimental): Early term (between 37 0/7 and 38 6/7 weeks)
  Interventions: Other: Early term group bathing 24 hours after birth.
- Group 4 (Experimental): Early term (between 37 0/7 and 38 6/7 weeks)
  Interventions: Other: Early term group bathing 48 hours after birth.

INTERVENTIONS:
Other: Preterm group bathing 24 hours after birth. — Preterm (between 32 0/7 and 36 6/7 weeks) babies (n=30) were bathed in the form of a shower 24 hours after birth. Before the bath, after the bath, 10 minutes after the bath and 60 minutes after the bath, heart rate, body temperature, respiratory rate, oxygen saturation value, and skin color were evaluated.
  Arms: Group 1
Other: Preterm group bathing 48 hours after birth. — Preterm (between 32 0/7 and 36 6/7 weeks) babies (n=30) were bathed in the form of a shower 48 hours after birth. Before the bath, after the bath, 10 minutes after the bath and 60 minutes after the bath, heart rate, body temperature, respiratory rate, oxygen saturation value, and skin color were evaluated.
  Arms: Group 2
Other: Early term group bathing 24 hours after birth. — Early term (between 37 0/7 and 38 6/7 weeks) babies (n=30) were bathed in the form of a shower 24 hours after birth. Before the bath, after the bath, 10 minutes after the bath and 60 minutes after the bath, heart rate, body temperature, respiratory rate, oxygen saturation value, and skin color were evaluated.
  Arms: Group 3
Other: Early term group bathing 48 hours after birth. — Early term (between 37 0/7 and 38 6/7 weeks) babies (n=30) were bathed in the form of a shower 48 hours after birth. Before the bath, after the bath, 10 minutes after the bath and 60 minutes after the bath, heart rate, body temperature, respiratory rate, oxygen saturation value, and skin color were evaluated.
  Arms: Group 4

SUMMARY:
The aim of this study is to examine the effect of the first bath timing after birth on the physiological variables of the newborn and to determine the correct bath time.

1. H₁: There is a difference in the effect of bathing preterm newborns after 24 hours or 48 hours on the peak heart rate.
2. H2: There is a difference in the effect of bathing early term newborns after 24 hours or 48 hours on the peak heart rate.
3. H3: There is a difference in the effect of bathing preterm newborns after 24 hours or 48 hours on their respiratory rate.
4. H4: There is a difference in the effect of bathing early term newborns after 24 hours or 48 hours on their respiratory rate.
5. H5: There is a difference in the effect of baths given to preterm newborns after 24 hours or 48 hours on body temperature.
6. H6: There is a difference in the effect of baths given to early term newborns after 24 hours or after 48 hours on body temperature.
7. H7: There is a difference in the effect of baths given to preterm newborns after 24 hours or 48 hours on oxygen saturation.
8. H8: There is a difference in the effect of baths given to early term newborns after 24 hours or after 48 hours on oxygen saturation.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of the first bath timing after birth on the physiological variables of the newborn and to determine the correct bath time. The research is a single-center, prospective parallel group randomized controlled experimental design study. The research was conducted with a total of 120 babies, 60 preterm babies and 60 early term babies, who received inpatient care and treatment in the neonatal intensive care unit between October 2022 and November 2023. Depending on randomization, newborns were bathed within 24 hours or 48 hours after birth. Physiological measurements of newborns were evaluated before application. Measurements were repeated after application, 10 minutes after application and 60 minutes after application. In the study, it was collected with the Baby Information Form and Physiological Variables Monitoring Form. Data were analyzed using chi-square, mean, percentage distributions, dependent groups t-test for comparison of intra-group measurements, repeated measures anova test, and independent groups t-test for comparison of quantitative continuous data. In the preterm group, the pre-bath respiration, body temperature and oxygen saturation values of newborns bathed within 48 hours were found to be significantly lower than those of newborns bathed within 24 hours in post-bath measurements (p<0.05). In the early term group, it was found that the pre-bath heart rate peak values of newborns bathed within 48 hours were significantly lower than those of newborns bathed within 24 hours in post-bath measurements (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Newborns should be between 32 0/7 and 38 6/7 weeks.
* Birth weight must be over 2000 grams.
* He should not be connected to a mechanical ventilator.
* The parent must agree to work.

Exclusion Criteria:

* Less than 32 0/7 weeks.
* 39 0/7 weeks over.
* Being connected to a mechanical ventilator.
* Lacking epidermal integrity.
* Having an infection.
* Babies with anomalies and syndromes.
* Whose mother has an infection (hepatitis B, hepatitis C, HIV).
* Having phototherapy treatment.
* Having a body temperature below 36.5 °C.
* Having a body temperature above 37.5 ºC.
* Feeding within an hour before bathing.
* A painful procedure is performed within thirty minutes before bathing.
* Taking sedative medication.
* Those whose parents do not allow them to work.

Ages: 32 Weeks to 38 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Body temperature | It was evaluated at 1 minute before bath, after bath, 10 minutes after bath and 60 minutes after bath.
  Body temperature will be recorded and evaluated in degrees Celsius.
Respiratory rate | It was evaluated at 1 minute before bath, after bath, 10 minutes after bath and 60 minutes after bath.
  Respiration will be recorded and evaluated in numbers by counting for 1 minute by the researcher.
Heart rate | It was evaluated at 1 minute before bath, after bath, 10 minutes after bath and 60 minutes after bath.
  Heart rate will be recorded and evaluated in numbers by measuring with a monitor,
Oxygen saturation value | It was evaluated at 1 minute before bath, after bath, 10 minutes after bath and 60 minutes after bath.
  Oxygen saturation value will be recorded and evaluated in numbers by the monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Health Application and Research Center Farabi Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.